CLINICAL TRIAL: NCT07003984
Title: A Phase 3 Global, Randomized, Double-Blind, Placebo-Controlled, Safety and Immunogenicity Study of CHIKV VLP Vaccine in Children 2 to <12 Years of Age
Brief Title: A Safety and Immunogenicity Study of CHIKV VLP Vaccine in Children.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EBSI-CV-317-006
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chikungunya Virus
Keywords: Chikungunya; PXVX0317; CHIKV VLP; vaccine; immunogenicity; VIMKUNYA; children
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by site and age subgroup, 6 to <12 years of age (Cohort 1) and 2 to <6 years of age (Cohort 2), and randomized in a 4:1 ratio to receive either a single intramuscular (IM) dose of 40 µg CHIKV VLP vaccine or placebo at Day 1. Using the same strata, participants will be randomized in a 1:1 ratio to attend Visit 2 at either Day 15 or Day 22.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Experimental): Cohort 1 Active Group
  Interventions: Biological: CHIKV VLP vaccine
- Arm 2 (Placebo Comparator): Cohort 1 Placebo Group
  Interventions: Biological: Placebo
- Arm 3 (Experimental): Cohort 2 Active Group
  Interventions: Biological: CHIKV VLP vaccine
- Arm 4 (Placebo Comparator): Cohort 2 Placebo Group
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CHIKV VLP vaccine — CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide (Alhydrogel®) adjuvant 2%
  Arms: Arm 1; Arm 3
Biological: Placebo — Placebo is comprised of formulation buffer
  Arms: Arm 2; Arm 4

SUMMARY:
The goal of this multi-center, randomized, double-blind, placebo-controlled study is to evaluate the safety and immunogenicity of CHIKV VLP Vaccine in children 2 to <12 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 2 and <12 years of age at Day 1 (day of vaccination).
2. In general good health, in the opinion of the investigator, based on medical history and physical examination.
3. Able and willing to provide informed assent for study participation and primary caregiver is able and willing to provide informed consent for study participation, in accordance with the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) determination and applicable federal and local regulations and guidelines.
4. Able and willing to complete all scheduled visits and comply with all study procedures.

Exclusion Criteria:

1. Participation or planned participation in an investigational clinical study (eg, vaccine, drug) within 30 days before Day 1 and for the duration of the study. Note: Participation in an observational study or follow-up phase of a study may be allowed; these instances should be discussed with the sponsor's medical monitor and written agreement obtained prior to enrollment.
2. Current acute illness, with or without fever.
3. Current or recent CHIKV infection indicated by positive immunoglobulin M (IgM) and negative immunoglobulin G (IgG) rapid diagnostic test (RDT) results at screening in the Philippines only; participants in the US will not be tested using the RDT.
4. History of any known or suspected allergy or history of anaphylaxis to any component of the investigational product.
5. History of any known congenital or acquired immunodeficiency or immunosuppressive condition that could impact response to vaccination.
6. Prior receipt or anticipated use of systemic immunomodulatory or immunosuppressive medications from 180 days prior to screening through Day 22. Note: Systemic corticosteroid use at a dose or equivalent dose of 20 mg or greater (≥0.5 mg/kg for children <40 kg) of prednisone for 14 consecutive days or more within 90 days of screening through Day 22 is exclusionary. The use of inhaled, intranasal, topical, or ocular steroids is allowed.
7. Receipt or anticipated receipt of immunoglobulin from 180 days prior to screening through the duration of the study.
8. Any administration or planned administration of:

   * A licensed live attenuated vaccine within 28 days before administration of investigational product and until Visit 2 (Day 15 or 22, as applicable) has occurred.
   * Other licensed (not live) vaccine within 14 days before administration of investigational product and until Visit 2 (Day 15 or 22, as applicable) has occurred.
   * Another licensed or investigational CHIKV vaccine.
9. Known infection with human immunodeficiency virus, hepatitis C virus (HCV), or hepatitis B virus. Note: Positive anti-HCV antibodies and negative HCV polymerase chain reaction would NOT be exclusionary. Polymerase chain reaction testing will not be performed as part of this protocol.
10. Bleeding disorder or receipt of anticoagulants in the 21 days before Day 1, contraindicating intramuscular vaccination, as judged by the investigator.
11. Receipt or anticipated receipt of blood products from 90 days before Day 1 through the duration of the study.
12. Onset of menarche prior to study vaccination.
13. Planned medical or surgical procedure that could adversely impact the participant's participation or the conduct of the study.
14. Identified as an immediate family member of the investigator or employee with direct involvement in the study. Bavarian Nordic staff members and their families, contractors, agents, business partners, and anyone with a financial interest in the outcome of the study.
15. Any other medical condition, including severe malnutrition, that, in the opinion of the investigator, could adversely impact the participant's participation or conduct of the study.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Primary Immunogenicity Endpoint: Day 22 anti-CHIKV SNA seroresponse rate in seronegative children | Study Day 22, 21 days after vaccination with CHIKV VLP vaccine or placebo.
  Day 22 anti-CHIKV serum neutralizing antibody (SNA) seroresponse rate in baseline seronegative children 2 to <12 years of age in the immunogenicity evaluable population.
Safety Endpoint 1: Incidence of solicited adverse events through Day 8 | From vaccination on study Day 1 through Day 8, 7 days after vaccination with CHIKV VLP vaccine or placebo.
  Incidence of solicited adverse events through Day 8.
Safety Endpoint 2: Incidence of unsolicited AEs through Day 29 | From vaccination on Day 1 through Day 29, 28 days after vaccination with CHIKV VLP vaccine or placebo.
  Incidence of unsolicited adverse events (AEs) through Day 29.
Safety Endpoint 3: Incidence of AESI, MAAEs, and SAEs | From vaccination through the end of the trial, planned to be Day 732 for study completers.
  Incidence of adverse events of special interest (AESIs; defined as new onset or worsening arthralgia that is medically attended), medically attended adverse events (MAAEs), and serious adverse events (SAEs) through end of the trial.

SECONDARY OUTCOMES:
Key Secondary Immunogenicity Endpoint 1: Day 15 anti-CHIKV SNA seroresponse rate in seronegative children | Study Day 15, 14 days after vaccination with CHIKV VLP vaccine or placebo.
  Day 15 anti-CHIKV serum neutralizing antibody (SNA) seroresponse rate in baseline seronegative children 2 to <12 years of age in the immunogenicity evaluable population.
Key Secondary Immunogenicity Endpoint 2: Day 22 anti-CHIKV SNA seroresponse rate in both seronegative and seropositive children | Study Day 22, 21 days after vaccination with CHIKV VLP vaccine or placebo.
  Day 22 anti-CHIKV serum neutralizing antibody (SNA) seroresponse rate in both baseline seronegative and seropositive children 2 to <12 years of age in the immunogenicity evaluable population.
Secondary Immunogenicity Endpoint 1: Day 15 anti-CHIKV SNA seroresponse rate in both seronegative and seropositive children | Study Day 15, 14 days after vaccination with CHIKV VLP vaccine or placebo.
  Day 15 anti-CHIKV serum neutralizing antibody (SNA) seroresponse rate in both baseline seronegative and seropositive children 2 to <12 years of age in the immunogenicity evaluable population.
Secondary Immunogenicity Endpoint 2: Day 183 and Day 366 anti-CHIKV SNA seroresponse rate in both seronegative and seropositive children | Study Day 183 and Day 366, 182 and 365 days after vaccination with CHIKV VLP vaccine or placebo, respectively.
  Day 183 and Day 366 anti-CHIKV serum neutralizing antibody (SNA) seroresponse rate in both baseline seronegative and seropositive children 2 to <12 years of age in the immunogenicity evaluable population.
Secondary Immunogenicity Endpoint 3: Day 15, Day 22, Day 183, and Day 366 anti-CHIKV SNA seroresponse rate in both seronegative and seropositive children | Day 15, Day 22, Day 183, and Day 366, 14, 21, 182, and 365 days after vaccination with CHIKV VLP vaccine or placebo, respectively.
  Day 15, Day 22, Day 183, and Day 366 anti-CHIKV serum neutralizing antibody (SNA) seroresponse rate in both baseline seronegative and seropositive children 2 to <12 years of age in the immunogenicity evaluable population, stratified by age stratum (2 to <6 and 6 to <12 years); analyzed by baseline serostatus separately and combined.
Secondary Immunogenicity Endpoint 4: GMTs of anti-CHIKV SNA at Day 15, Day 22, Day 183, and Day 366 for the CHIKV VLP vaccine and placebo groups, and Day 732 for CHIKV VLP vaccine group only | Day 15, Day 22, Day 183, Day 366, and Day 732, 14, 21, 182, 365, and 731 days after vaccination, respectively.
  Geometric mean titers (GMTs) of anti-CHIKV serum neutralizing antibodies (SNA) at Day 15, Day 22, Day 183, and Day 366 for the CHIKV VLP vaccine and placebo groups, and Day 732 for CHIKV VLP vaccine group only, in children 2 to <12 years of age in the immunogenicity evaluable population by age stratum (2 to <6 and 6 to <12 years); analyzed by baseline serostatus separately and combined.
Secondary Immunogenicity Endpoint 5a: GMFIs from Day 1 to Day 15, Day 22, Day 183, and Day 366 for the CHIKV VLP vaccine and placebo groups, and Day 732 for CHIKV VLP vaccine group only | Day 15, Day 22, Day 183, Day 366, and Day 732, 14, 21, 182, 365, and 731 days after vaccination, respectively.
  Geometric mean fold increases (GMFIs) from Day 1 (prevaccination) to Day 15, Day 22, Day 183, and Day 366 for the CHIKV VLP vaccine and placebo groups, and Day 732 for CHIKV VLP vaccine group only in children 2 to <12 years of age in the IEP and by age stratum (2 to <6 and 6 to <12 years); analyzed by baseline serostatus separately and combined.
Secondary Immunogenicity Endpoint 5b: Frequency of participants with titer ≥15 and 4-fold rise over baseline at Day 15, Day 22, Day 183, and Day 366 for the CHIKV VLP vaccine and placebo groups, and Day 732 for the CHIKV VLP vaccine group only | Day 15, Day 22, Day 183, Day 366, and Day 732, 14, 21, 182, 365, and 731 days after vaccination, respectively.
  Frequency of participants with titer ≥15 and 4-fold rise over baseline at Day 15, Day 22, Day 183, and Day 366 for the CHIKV VLP vaccine and placebo groups, and Day 732 for the CHIKV VLP vaccine group only in children 2 to <12 years of age in the IEP and by age stratum (2 to <6 and 6 to <12 years); analyzed by baseline serostatus separately and combined.
Secondary Immunogenicity Endpoint 6: Anti-CHIKV SNA seroresponse rates at Day 732 in the CHIKV VLP vaccine group only | Study Day 732, 731 days after vaccination with CHIKV VLP vaccine.
  For the CHIKV VLP vaccine group only, anti-CHIKV serum neutralizing antibody (SNA) seroresponse rates at Day 732 in both baseline seronegative and seropositive children 2 to <12 years of age and by age stratum (2 to <6 and 6 to <12 years); analyzed by baseline serostatus separately and combined.
Secondary Immunogenicity Endpoint 7: Day 22 anti-CHIKV SNA seroresponse rate between seronegative children in the IEP versus adolescents and adults study EBSI-CV-317-004 | Study Day 22, 21 days after vaccination with CHIKV VLP vaccine or placebo.
  Day 22 anti-CHIKV serum neutralizing antibody (SNA) seroresponse rate between baseline seronegative children 2 to <12 years of age in the immunogenicity evaluable population (IEP) versus adolescents and adults from 12 to <65 years of age in study EBSI-CV-317-004.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ajiboye, MD, Study Director — Bavarian Nordic A/S
Locations (9):
- United States (8):
  - ARK Clinical Research, LLC, Fountain Valley, California
  - Emerson Clinical Research Institute- DC, Washington D.C., District of Columbia
  - Acevedo Clinical Research, Miami, Florida
  - Hope Research Network, Miami, Florida
  - Velocity Clinical Research-Omaha, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - KidCare Pediatrics, Beaumont, Texas
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
- Caribbean Medicine Center, San Juan, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett SR, McCarty JM, Ramanathan R, Mendy J, Richardson JS, Smith J, Alexander J, Ledgerwood JE, de Lame PA, Royalty Tredo S, Warfield KL, Bedell L. Safety and immunogenicity of PXVX0317, an aluminium hydroxide-adjuvanted chikungunya virus-like particle vaccine: a randomised, double-blind, parallel-group, phase 2 trial. Lancet Infect Dis. 2022 Sep;22(9):1343-1355. doi: 10.1016/S1473-3099(22)00226-2. Epub 2022 Jun 13. PMID 35709798
- [Background] McCarty JM, Bedell L, Mendy J, Coates EE, Chen GL, Ledgerwood JE, Tredo SR, Warfield KL, Richardson JS. Chikungunya virus virus-like particle vaccine is well tolerated and immunogenic in chikungunya seropositive individuals. Vaccine. 2023 Oct 6;41(42):6146-6149. doi: 10.1016/j.vaccine.2023.08.086. Epub 2023 Sep 9. PMID 37690874
- [Background] Richardson JS, Anderson DM, Mendy J, Tindale LC, Muhammad S, Loreth T, Tredo SR, Warfield KL, Ramanathan R, Caso JT, Jenkins VA, Ajiboye P, Bedell L; EBSI-CV-317-004 Study Group. Chikungunya virus virus-like particle vaccine safety and immunogenicity in adolescents and adults in the USA: a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2025 Apr 19;405(10487):1343-1352. doi: 10.1016/S0140-6736(25)00345-9. Epub 2025 Mar 27. PMID 40158526